CLINICAL TRIAL: NCT02031601
Title: Randomised, Controlled Study Comparing Chemotherapy Plus Intercalated EGFR-Tyrosine Kinase Inhibitors Combination Therapy With EGFR-Tyrosine Kinase Inhibitors Alone Therapy as First-line Treatment for Patients With Non-Small-Cell Lung Cancer
Brief Title: Intercalated Combination of Chemotherapy and Tyrosine Kinase Inhibitors as First-line Treatment for Patients With Non-Small-Cell Lung Cancer
Acronym: TCL-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qian Qi, assistant director, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLHX-0531
Record Dates: First submitted 2014-01-02; First posted 2014-01-09 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2015-11

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gefitinib; icotinib; Docetaxel; Pemetrexed; Platinum; Cisplatin; Carboplatin

ARMS (2):
- Combination therapy (Experimental): Interventions:
  Drug: Erlotinib [Tarceva] or Gefitinib [Iressa] or Icotinib [Conmana] plus Drug: Docetaxel for patients of lung squamous cell carcinoma; Pemetrexed for patients of lung adenocarcinoma plus Drug: Platinum (cisplatin or carboplatin)
  Interventions: Drug: Erlotinib; Drug: Gefitinib; Drug: Icotinib; Drug: Docetaxel; Drug: Pemetrexed; Drug: Platinum (cisplatin or carboplatin)
- TKI alone therapy (Other): Interventions:
  Drug: Erlotinib [Tarceva] or Gefitinib [Iressa] or Icotinib [Conmana]
  Interventions: Drug: Erlotinib; Drug: Gefitinib; Drug: Icotinib

INTERVENTIONS:
Drug: Erlotinib — 150mg po once a day on days 2-15 of each 3 week cycle for 4 cycles; then continue to receive erlotinib150mg po once a day daily until progression
  Other Names: Tarceva
  Arms: Combination therapy
Drug: Gefitinib — 250mg po once a day on days 2-15 of each 3 week cycle for 4 cycles; then continue to receive gefitinib 250mg po once a day daily until progression
  Other Names: Iressa
  Arms: Combination therapy
Drug: Icotinib — 125mg po three time a day on days 2-15 of each 3 week cycle for 4 cycles; then continue to receive icotinib 125mg po three time a day daily until progression
  Other Names: Conmana
  Arms: Combination therapy
Drug: Docetaxel — 75 mg/m2 ivgtt on days 1 of each 3 week cycle for 4 cycles
  Arms: Combination therapy
Drug: Pemetrexed — 500 mg/m2 ivgtt on days 1 of each 3 week cycle for 4 cycles
  Arms: Combination therapy
Drug: Platinum (cisplatin or carboplatin) — cisplatin -- 75mg/m2 ivgtt on day 1 of each 3 week cycle for 4 cycles or carboplatin -- 5 x AUC ivgtt on day 1 of each 3 week cycle for 4 cycles
  Arms: Combination therapy
Drug: Erlotinib — 150mg po once a day daily until disease progression
  Other Names: Tarceva
  Arms: TKI alone therapy
Drug: Gefitinib — 250mg po once a day daily until disease progression
  Other Names: Iressa
  Arms: TKI alone therapy
Drug: Icotinib — 125mg po three times a day daily until disease progression
  Other Names: Conmana
  Arms: TKI alone therapy

SUMMARY:
Objective: To compare the efficacy and safety of chemotherapy plus intercalated EGFR-tyrosine kinase inhibitors (TKI) combination therapy with TKI alone therapy as first-line treatment for patients with non-small-cell lung cancer (NSCLC).

Methods: Patients with untreated, stage IIIB/IV, EGFR mutation-positive NSCLC will be randomly assigned to combination therapy group (receiving four cycles of docetaxel or pemetrexed (on day 1) plus platinum (on day 1) with intercalated TKI (gefitinib, erlotinib or Icotinib, on day 2-15) every 3 weeks) or TKI alone therapy (gefitinib, erlotinib or Icotinib, daily). All patients were continued to receive TKI until progression or unacceptable to toxicity or death. The primary endpoint was progression-free survivial (PFS).

Expected results: PFS of combination therapy group will be prolonged to nineteen months while PFS of TKI alone therapy group is ten months. Overall survival (OS) of combination therapy group will be prolonged to 36 months while OS of TKI alone therapy group is 26 months.

Hypothesis: Platinum-based chemotherapy plus intercalated TKI combination therapy as first-line treatment will prolong PFS and OS for patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age;
* Advanced (stage IIIB/IV) non-small-cell lung cancer;
* Although stageⅠ-ⅢA, have contraindications to surgery;
* EGFR mutation-positive (EGFR exon-18, exon-19 or exon-21);
* Measurable disease;
* ECOG Performance Status 0 or 1 or 2.

Exclusion Criteria:

* Wild-type EGFR;
* Prior exposure to agents directed at the HER axis;
* Prior chemotherapy or systemic anti-tumor therapy after advanced disease;
* Unstable systemic disease;
* Any other malignancy within last 5 years, except cured basal cell cancer of skin or cured cancer in situ of cervix;
* Brain metastasis or spinal cord compression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 8 weeks
  Progression-free survival (PFS) is defined to be the time from randomization to progression of disease or death, whichever occurs first. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study, or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
Objective response rate | 8 weeks
Duration of response | 8 weeks
Time to progression | 8 weeks
Overall survival (OS) | 8 weeks
Clinical benefit rate | 8 weeks
Adverse Events (AEs), Serious Adverse Events (SAEs), laboratory data | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu Li, Professor, Study Director — Director
Locations (1):
- Yu Li, Jinan, Shandong, China

REFERENCES:
- [Derived] Xu L, Qi Q, Zhang Y, Cui J, Liu R, Li Y. Combination of icotinib and chemotherapy as first-line treatment for advanced lung adenocarcinoma in patients with sensitive EGFR mutations: A randomized controlled study. Lung Cancer. 2019 Jul;133:23-31. doi: 10.1016/j.lungcan.2019.05.008. Epub 2019 May 7. PMID 31200823